CLINICAL TRIAL: NCT07334418
Title: EAGLET-CS Pilot: Early General Anesthesia to Limit Experiences of Trauma During Cesarean Section-Pilot Study
Brief Title: Early General Anesthesia to Limit Experiences of Trauma During Cesarean Section-Pilot Study
Acronym: EAGLET-CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Mark Neuman, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 859498
Record Dates: First submitted 2025-12-02; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section; Delivery; Trauma
Keywords: Cesarean Section; Delivery; Trauma; C-section; PTSD
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Anesthetics, General; Anesthetics, Intravenous

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Comparator 1: Standard-care general anesthesia: medically induced unconsciousness with breathing tube placement.
  Interventions: Drug: General anesthetic
- Intravenous sedation (Active Comparator): Comparator 2: Time-limited trial of standard care minimal-to-moderate intravenous sedation, with conversion to general anesthesia if pain persists.
  Interventions: Drug: Intravenous anesthetic

INTERVENTIONS:
Drug: General anesthetic — standard of care general anesthesia
  Arms: General anesthesia
Drug: Intravenous anesthetic — standard of care intravenous anesthesia
  Arms: Intravenous sedation

SUMMARY:
Some patients who undergo cesarean section under spinal or epidural anesthesia can experience severe pain. Some patients who experience this kind of pain can experience symptoms of post-traumatic stress disorder (PTSD) after pregnancy. Currently, the two main options for treating this pain are general anesthesia (full medically induced unconsciousness) and using intravenous medications to reduce the pain and decrease anxiety. The EAGLET-CS Pilot is a pilot randomized trial that will test the feasibility of comparing the impact of these two options for preventing PTSD in a rigorous way for those patients who experience pain during their cesarean section after the baby is out.

DETAILED DESCRIPTION:
The EAGLET-CS Pilot is a randomized trial that will assess the feasibility of comparing two commonly used approaches to care for women undergoing cesarean delivery under standard neuraxial anesthesia (epidural, spinal, or CSE) who experience intraoperative pain after delivery that is refractory to first line treatments. 12 patients recruited from the labor and delivery service at the Hospital of the University of Pennsylvania will be assigned to one of two standard-care comparators, namely early conversion to general anesthesia versus a time-limited trial of intravenous sedation, followed by conversion to general anesthesia if needed due to ongoing pain. Patients will be assessed during hospitalization and at up to 6 weeks after delivery to assess mental health, medical, and quality of recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older undergoing non-emergent cesarean delivery with primary neuraxial (epidural, spinal, or CSE) anesthesia. Eligible patients will be those who report severe pain during surgery, defined as pain that does not resolve with 2 trials of first-line pharmacologic therapies (e.g., epidural supplementation with local anesthetics; intravenous opioid analgesics).

Exclusion Criteria:

* We will exclude patients who require induction of general anesthesia prior to umbilical cord clamping and by clinician determination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Consent | From hospital admission through day of delivery
  Study consent rate, defined as the number of patients consenting to participation among those approached for enrollment.

SECONDARY OUTCOMES:
Percentage of patients meeting all inclusion criteria out of all screened | From hospital admission through day of delivery
  Percentage of patients meeting all inclusion criteria out of all screened
Randomization | From hospital admission through day of delivery
  Percentage of consenting patients who undergo study randomization
Quality of postoperative recovery | Postoperative day 0, 1, 2, or 3
  Quality of postoperative recovery via 11-item Obstetric Quality of Recovery Scoring Tool minimum score 0 and maximum score 110. A higher score means better.
Satifaction with anesthesia | Postoperative day 0, 1, 2, or 3
  Satisfaction with anesthesia care via 11-item Obstetric Quality of Recovery Scoring Tool minimum score 0 and maximum score 110. A higher score means better.
Severity and duration of pain | Postoperative day 0, 1, 2, or 3
  Reported severity and duration of pain during surgery via 5-item SONAR (Snapshot Obstetric Anesthesia National Research Project) Maternal Comfort Scale. Minimum score 5 and Maximum score 35. A higher score means better.
Adverse events | Randomization through postoperative day 30
  Postoperative serious adverse events via chart review
Length of stay | Randomization through postoperative day 30
  Post-randomization hospital length of stay via chart review
Need for intensive care | Randomization through postoperative day 30
  Need for maternal intensive care via chart review
New PTSD (Posttraumatic Stress Disorder) symptoms | Postoperative 6 week
  New PTSD (Posttraumatic Stress Disorder) symptoms at 6 weeks after delivery via PCL-5 (Posttraumatic Stress Disorder Checklist for DSM-5) Minimum score 0 and maximum score 80. A higher score means worse.

IPD SHARING:
Plan to Share IPD: No